CLINICAL TRIAL: NCT03072277
Title: Maternal Docosa-Hexaenoic Acid (DHA) Supplementation and Offspring Neurodevelopment in India (DHANI-2)
Brief Title: Maternal DHA Supplementation and Offspring Neurodevelopment in India (DHANI-2)
Acronym: DHANI-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Public Health Foundation of India (Other)
Collaborators: Jawaharlal Nehru Medical College (Other); India Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IA/CPHE/14/1/501498
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy
Keywords: DHA; Docosa Hexaenoic Acid; Omega 3 fatty acid; Birth Outcome; Birth Size; Gestational Age; DASII; Prenatal and Postnatal Supplementation; Randomized Controlled Trial; Neurodevelopment; Pregnancy; Lactation
MeSH Terms: conditions — Breast Feeding | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, parallel arm hospital based trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docosa Hexaenoic Acid (DHA) (Active Comparator): Omega 3 Fatty Acid
  Interventions: Dietary Supplement: Docosa Hexaenoic Acid (DHA)
- Placebo (Placebo Comparator): Corn/Soy Oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosa Hexaenoic Acid (DHA) — 400 mg/day of Docosa-hexaenoic Acid (algal DHA) will given to the pregnant women (in the active group) from ≤20 weeks of gestation through 6 months postpartum.
  Other Names: Omega 3 Fatty Acid
  Arms: Docosa Hexaenoic Acid (DHA)
Dietary Supplement: Placebo — 400 mg/day of placebo (corn/soy oil) will be given to the pregnant women from ≤20 weeks of gestation through 6 months postpartum.
  Other Names: Corn/Soy oil
  Arms: Placebo

SUMMARY:
DHANI-2 is an extension to DHANI (NCT01580345) which proposes to extend maternal supplementation (DHA or Placebo) from <20 weeks of gestational age through 6 months postpartum and infant follow-up through 12 months. Leveraging the Randomized Controlled Trial (RCT) design, DHANI-2 aims to assess the role of maternal DHA supplementation on infant neurodevelopment and body growth. It also intends to enhance the mechanistic understanding by the addition of repeated biochemical measures from mother-child dyads.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo controlled trial would be conducted among pregnant women in India to test the effectiveness of supplementing pregnant Indian women with 400 mg/d algal DHA compared to placebo from mid-pregnancy through delivery. Eligible participants would be randomized to receive either 400 mg of DHA or a placebo baseline measures would be taken before the enrollment of the participant in the study. The mother-child dyads would be followed through infant age 1 year and anthropometric measurements and biochemical investigations would be used to assess the effect of maternal DHA supplementation on infant neurodevelopment at ages 6- and 12-months using validated the Development Assessment Scale for Indian Infants (DASII).

ELIGIBILITY:
Inclusion Criteria:

* Willing, healthy singleton gestation of ≤ 20 weeks (scan report must)
* 18-35 years
* Hb > 7 g/dL
* Non-fasting glucose as per Diabetes in Pregnancy Study Group of India (DIPSI) criteria (<140mg/dL)
* No history of chronic diseases (heart disease, diabetes, liver disorders, cancer, epilepsy, HIV, thyroid) or
* High risk pregnancy (short stature**, molar pregnancy++, HBsAg positive, as advised by physicians)

  * <143 cm ++ A molar pregnancy starts when an egg is fertilized, but instead of a normal, viable pregnancy resulting, the placenta develops into an abnormal mass of cysts.

Exclusion Criteria:

* Women allergic (if aware) to any of the test products.
* Women at high risk for hemorrhagic bleeding, clotting (if aware).
* Women with high-risk pregnancies (history and prevalence of pregnancy complications, including abruptio placentae, preeclampsia, pregnancy-induced hypertension, any serious bleeding episode in the current pregnancy, and/ or physician referral); and/or diagnosed chronic degenerative disease(s) such as diagnosed heart disease, cancer, stroke or diabetes (as omega-3 could raise blood sugar and lower insulin production).
* Women consuming omega-3 supplements or having used these in 3 months preceding the intervention period.
* Reported participation in another biomedical trial 3 months before the start of the study or during the study (not to get the results of the present study contaminated).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 957 (Actual)
Dates: Start 2015-12; Primary Completion 2019-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Infant neurodevelopment as measured by his/her Development quotient scores (DQS) at 12 months of age | 12 months (± 4 weeks)
  The development quotient (DQ) among infants at 12 months of age assessed using the standardized Development Assessment Scale for Indian Infants (DASII). DASII is the Indian modification (done in 1970 and 1977) of the Bayley Scale of Infant Development (BSID) using Indian norms for 67 motor and 163 mental items of the BSID. DASII provides a measure of DQ among Indian infants below 30 months of age. DQ is defined as the ratio of functional to chronological age. Third, 50th and 97th percentile norms are given. A higher score indicates a better outcome. The maximum DQ score is 100; ≥85 is normal; 71-84 is mild to moderate delay and developmental delay is defined as DQ ≤70 (≤2SD). Median reliability index for motor and mental scales based on correlation between consecutive months is noted to be 0.88 for motor scales and 0.91 for mental scales.

SECONDARY OUTCOMES:
Mean difference in infant developmental quotient (DQ) at 6 month | 6 months (± 4 weeks)
  Mean Difference in the infant developmental quotient (DQ) as measured by the Development Assessment Scale for Indian Infants (DASII) at 6 months. DASII is the Indian modification (done in 1970 and 1977) of the Bayley Scale of Infant Development (BSID) using Indian norms for 67 motor and 163 mental items of the BSID. DASII provides a measure of DQ among Indian infants below 30 months of age. DQ is defined as the ratio of functional to chronological age. Third, 50th and 97th percentile norms are given. A higher score indicates a better outcome. The maximum DQ score is 100; ≥85 is normal; 71-84 is mild to moderate delay and developmental delay is defined as DQ ≤70 (≤2SD).
Mean difference in infant motor score at 6 month | 6 (± 4 weeks)
  Mean Difference in the motor score as measured by the Development Assessment Scale for Indian Infants (DASII) at 6 months. DASII is the Indian modification (done in 1970 and 1977) of the Bayley Scale of Infant Development (BSID) using Indian norms for 67 motor and 163 mental items of the BSID. A higher score indicates a better outcome. The motor development items cover the child's development from supine to erect posture, neck-control, locomotion etc. It also includes the record for manipulative behaviour such as reaching, picking-up, handling things etc.
Mean difference in infant mental score at 6 month | 6 months (± 4 weeks)
  Mean Difference in the mental score as measured by the Development Assessment Scale for Indian Infants (DASII) at 6 months. DASII is the Indian modification (done in 1970 and 1977) of the Bayley Scale of Infant Development (BSID) using Indian norms for 67 motor and 163 mental items of the BSID. A higher score indicates a better outcome. The mental development items record the child's cognizance of objects in the surroundings, perceptual pursuit of moving objects, exploring them to meaningful manipulation. It also covers the development of communication and language comprehension, spatial relationship and manual dexterity, imitative behavior and social interaction etc.
Difference in numbers / proportions of infants with developmental delay | 6 months (± 4 weeks) and 12 (± 4 weeks) months
  Difference in numbers / proportions of infants with developmental delay between the Docosa-hexaenoic acid (DHA) and placebo group at 6 and 12 months. Developmental delay will be defined as a Development Quotient score ≤70 as assessed by Development Assessment Scale for Indian Infants (DASII).
Mean difference in infant weight (in grams) at birth | At delivery
  Mean difference in infant weight score between the Docosahexaenoic acid (DHA) and placebo group at birth. Birth weight is measured to the nearest 10 g by using a digital pediatric scale. Low birth weight is defined as recorded birth weight less than 2500 g.
Mean difference in infant (in centimeters) at birth | At delivery
  Mean difference in infant length between the Docosahexaenoic acid (DHA) and placebo group at birth. Birth length is the height of infant from maximum convexity of head to heel of the foot of the baby just after birth. It is measured using a portable infantometer with a fixed headpiece according to standard procedures. The Body length at birth is recorded in centimetres (cm) to 1 decimal place.
Mean difference in infant head circumference (in centimeters) at birth | At delivery
  Mean difference in infant head circumference between the Docosahexaenoic acid (DHA) and placebo group at birth. Birth length is the measurement of a child's head around its largest area - the distance from above the eyebrows and ears and around the back of the head. It is measured using non-stretchable measuring tape. It should be written in cm to 1 decimal place.
Mean difference in infant APGAR (Appearance, Pulse, Grimace, Activity, Respiration) score at birth. | At delivery
  Mean difference in APGAR (Appearance, Pulse, Grimace, Activity, Respiration) score between the Docosahexaenoic acid (DHA) and placebo group at birth. The APGAR score is a way to quickly measure and simply the health of an infant immediately after birth by adding the scores of the five criteria- Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability/ response), Activity (muscle tone) and Respiration to come up with a single number. This test is done at 1, 5 minutes. A low score on the 1-minute test may show that the neonate requires medical attention but is not necessarily an indication that there will be long-term problem.
Mean change in infant weight (in grams) at birth, 1 month, 6 months and 12 months between the Docosahexaenoic acid (DHA) and placebo group | At delivery, 1 month (± 4 weeks), 6 months (± 4 weeks) and, 12 months (± 4 weeks)
  Mean change in infant weight at birth, 1 month, 6 months and 12 months between the Docosahexaenoic acid (DHA) and placebo group. Birth weight is measured to the nearest 10 g by using a digital pediatric scale. Low birth weight is defined as recorded birth weight less than 2500 g.
Mean change in infant length (in centimeters) at birth, 1 month, 6 months and 12 months between the Docosahexaenoic acid (DHA) and placebo group | At delivery, 1 month (± 4 weeks), 6 months (± 4 weeks) and, 12 months (± 4 weeks)
  Mean change in infant length Docosahexaenoic acid (DHA) and placebo group at birth, 1 month, 6 months and 12 months between the DHA and placebo group. Birth length is the height of infant from maximum convexity of head to heel of the foot of the baby just after birth. It is measured using a portable infantometer with a fixed headpiece according to standard procedures. The Body length at birth is recorded in centimetres (cm) to 1 decimal place.
Mean change in infant head circumference (in centimeters) at birth, 1 month, 6 months and 12 months between the Docosahexaenoic acid (DHA) and placebo group | At delivery, 1 month (± 4 weeks), 6 months (± 4 weeks) and, 12 months (± 4 weeks)
  Mean change in infant size head circumference Docosahexaenoic acid (DHA) and placebo group at birth, 1 month, 6 months and 12 months between the Docosahexaenoic acid (DHA) and placebo group. Mean difference in infant head circumference between the Docosahexaenoic acid (DHA) and placebo group at birth. Birth length is the measurement of a child's head around its largest area - the distance from above the eyebrows and ears and around the back of the head. It is measured using non-stretchable measuring tape. It should be written in cm to 1 decimal place.
Mean difference in proportions of still births between Docosahexaenoic acid (DHA) and placebo groups. | At delivery
  Mean difference in proportions of still births between Docosahexaenoic acid (DHA) and placebo groups. Stillbirths are defined as fetuses delivered at 20 weeks of gestation or later with no signs of life and recorded as occurring before or during the onset of labor.
Mean difference in proportions of preterm babies between Docosahexaenoic acid (DHA) and placebo groups. | At delivery
  Mean difference in proportions of preterm babies between Docosahexaenoic acid (DHA) and placebo groups. Preterm delivery is defined as delivery after 20 weeks and before 37 weeks of completed gestation. Foetal losses during pregnancy - including miscarriages/abortions and still-births are recorded by study personnel on site or details are brought by field workers (in case mother went to any other hospital).
Mean difference in proportions of low birth weight babies between Docosahexaenoic acid (DHA) and placebo groups. | At delivery
  Mean difference in proportions of low birth weight babies between Docosahexaenoic acid (DHA) and placebo groups. Low birth weight is defined as recorded birth weight less than 2500 g.
Difference in infant morbidity patterns between Docosahexaenoic acid (DHA) and placebo groups | 1 month (± 4 weeks), 6 months (± 4 weeks) and, 12 months (± 4 weeks)
  Difference in infant morbidity patterns (types of illness, frequency and duration of specific conditions) between DHA and placebo group. Information collected on infant morbidity include questions reporting of illnesses - cough, nasal congestion, difficulty in breathing, cyanosis, convulsions, fever, vomiting, rash, ear discharge, excessive crying, and diarrhoea from birth till the age of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- KLEUs Jawaharlal Nehru Medical College -- Prabhakar Kore Charitable Hospital, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khandelwal S, Swamy MK, Patil K, Kondal D, Chaudhry M, Gupta R, Divan G, Kamate M, Ramakrishnan L, Bellad MB, Gan A, Kodkany BS, Martorell R, Srinath Reddy K, Prabhakaran D, Ramakrishnan U, Tandon N, Stein AD. The impact of DocosaHexaenoic Acid supplementation during pregnancy and lactation on Neurodevelopment of the offspring in India (DHANI): trial protocol. BMC Pediatr. 2018 Aug 4;18(1):261. doi: 10.1186/s12887-018-1225-5. PMID 30077178
- [Result] Khandelwal S, Kondal D, Chaudhry M, Patil K, Swamy MK, Metgud D, Jogalekar S, Kamate M, Divan G, Gupta R, Prabhakaran D, Tandon N, Ramakrishnan U, Stein AD. Effect of Maternal Docosahexaenoic Acid (DHA) Supplementation on Offspring Neurodevelopment at 12 Months in India: A Randomized Controlled Trial. Nutrients. 2020 Oct 3;12(10):3041. doi: 10.3390/nu12103041. PMID 33023067
- [Result] Khandelwal S, Kondal D, Chaudhry M, Patil K, Swamy MK, Pujeri G, Mane SB, Kudachi Y, Gupta R, Ramakrishnan U, Stein AD, Prabhakaran D, Tandon N. Prenatal Maternal Docosahexaenoic Acid (DHA) Supplementation and Newborn Anthropometry in India: Findings from DHANI. Nutrients. 2021 Feb 25;13(3):730. doi: 10.3390/nu13030730. PMID 33668849
- See also: The impact of DocosaHexaenoic Acid supplementation during pregnancy and lactation on Neurodevelopment of the offspring in India (DHANI): trial protocol — https://pubmed.ncbi.nlm.nih.gov/30077178/
- See also: Effect of Maternal Docosahexaenoic Acid (DHA) Supplementation on Offspring Neurodevelopment at 12 Months in India: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/33023067/
- See also: Prenatal Maternal Docosahexaenoic Acid (DHA) Supplementation and Newborn Anthropometry in India: Findings from DHANI — https://pubmed.ncbi.nlm.nih.gov/33668849/